CLINICAL TRIAL: NCT02917005
Title: A Phase II Study of Ovarian Function Suppression And ExemesTane With or Without PalbocIclib in PreMenopausal Women With ER Positive / HER-2 Negative MetAstatic Breast Cancer
Brief Title: PalbocIclib in PreMenopausal Women With ER Positive/HER-2 Negative MetAstatic Breast Cancer
Acronym: FATIMA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamdy A. Azim (Other)
Responsible Party: Sponsor-Investigator, Hamdy A. Azim, Prof, Africa Middle East Cancer Intergroup
Organization: Africa Middle East Cancer Intergroup (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMCI-001
Record Dates: First submitted 2016-09-18; First posted 2016-09-28 (Estimated); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Metastatic Breast Cancer
Keywords: breast cancer; hormone receptor positive, HER2 negative; palbociclib; premenopausal
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib; exemestane; Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Palbociclib Arm (Experimental): Palbociclib (Pfizer) 125mg/day orally for 3 weeks followed by 1 week off plus Exemestane (Pfizer) 25mg/day orally continuously plus Goserelin (Astrazeneca) 3.6 mg SC given every 28 days
  Interventions: Drug: Palbociclib; Drug: Exemestane; Drug: Goserelin
- Control Arm (Active Comparator): Exemestane (Pfizer) 25mg/day orally continuously plus Goserelin (Astrazeneca) 3.6 mg SC given every 28 days
  Interventions: Drug: Exemestane; Drug: Goserelin

INTERVENTIONS:
Drug: Palbociclib — CDK 4/6 inhibitor
  Other Names: Ibrance
  Arms: Palbociclib Arm
Drug: Exemestane — Aromatase inhibitor
  Other Names: Aromasine
Drug: Goserelin — LHRH agonist
  Other Names: Zoladex

SUMMARY:
This is an open label, randomized, multicenter, international phase II study for premenopausal patients with hormone receptor positive, HER2 negative metastatic or locally advanced breast cancer. Patients will be randomized to receive either palbociclib + exemestane + OFS (Arm 1) or exemestane +OFS (Arm 2).

Treatment will be continued until disease progression, unacceptable toxicities, or withdrawal of consent.

DETAILED DESCRIPTION:
There is a strong in-vitro and clinical evidence suggesting that the dual inhibition of CDK 4/6 and ER signaling is a highly effective therapeutic strategy in HR+ MBC. With the unprecedented success of palbociclib in PALOMA-1 trial, several phase 2 and 3 trials are underway to evaluate this agent (and other CDK4/6 inhibitors as well) in the different clinical scenarios of HR+ breast cancer [28].The vast majority of these trials -if not all- are testing these novel agents in postmenopausal patients, which would render the clinical experience of these agents restricted to postmenopausal women (median age was 62 years in PALOMA-1 trial) The scarcity of clinical trials addressing endocrinal therapy in premenopausal women with MBC is, at least in part, related to the fact that the majority of women in western countries are diagnosed with breast cancer during their postmenopausal life. However the situation is rather different in many countries, including those in the Middle East region, where the median age of women diagnosed with breast cancer is below 50 years, and where approximately 50% of these patients are still menstruating.

This study will be the first to explore the therapeutic effects of palbociclib when combined with exemestane and ovarian function suppression (OFS) in premenopausal with hormone receptor positive and HER2 negative MBC, and how it will compare to the classic approach of using OFS plus an aromatase inhibitor.

ELIGIBILITY:
Inclusion Criteria:

1. Adult women (≥ 18 years of age) with metastatic or locally advanced breast cancer (histologically or cytologically proven diagnosis of adenocarcinoma of the breast) not amenable to curative treatment by surgery or radiotherapy.
2. ER positive tumour: Histological or cytological confirmation of estrogen and/or progesterone-receptor positive, as determined by routine IHC. Positivity is defined as ≥1% positive stained cells. The receptor status determined by utilizing an assay consistent with local laboratory standards.
3. HER2 negative breast cancer as confirmed by IHC, SISH or FISH.
4. Premenopausal women : (definition of a real menopause is not a simple task in these relatively young women, owing to the potential effect of prior chemotherapy and /or endocrinal therapy particularly OFS) defined either by:

   i. Any age below 40 years , irrespective to E2 level or menstrual history ii. If the woman had a menstrual period any time within the last 12 months iii. If the woman has amenorrhea of more than 12 months (in the absence of chemotherapy or ovarian function suppression) that is associated with serum hormone levels that are NOT in the postmenopausal range (either estradiol (E2) < 30 pg/mL and follicle-stimulating hormone (FSH) < 20 mU/mL OR E2 ≥ 30 pg/mL and FSH ≥ 20 mU/mL) [30].
5. Secondary hormonal resistance to tamoxifen or endocrinal sensitive metastatic disease i. Secondary hormonal resistance is defined as recurrence after 24 months from the start of adjuvant tamoxifen treatment or within 12 months from the end of the 5 years of adjuvant Tamoxifen ii. Endocrinal sensitive disease is defined as recurrence after 12 months from the end of adjuvant tamoxifen treatment or de novo metastatic disease
6. Measurable disease according to RECIST or bone-only metastases. Previously irradiated lesions are deemed measurable only if progression is documented at the site after completion of radiation.

   i. Patients must either have at least one lesion that can be accurately measured; OR ii. Patients have bone lesions: lytic or mixed (lytic + sclerotic) in the absence of measurable disease as defined above.
7. ECOG Performance Status 0, 1, & 2.
8. Resolution of all acute toxic effects of prior therapy or surgical procedures to National Cancer Institute (NCI) CTCAE Grade 1 (except alopecia or other toxicities not considered a safety risk for the patient).
9. Adequate organ function as defined by the following criteria:

   i. Absolute neutrophil count (ANC) ≥ 1.5 10˄9/L ii. Platelets > 100 x10˄9/L iii. Hemoglobin (Hgb) > 9.0g/dL iv. INR < 2 v. Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.5x ULN (or <5 if hepatic metastases are present) vi. Total serum bilirubin < 1.5 x ULN (<3 x ULN for patients known to have Gilberts Syndrome) vii. Serum creatinine < 1.5 x ULN viii. QTc< 470 msec (based on the mean value of the triplicate ECGs).
10. Written informed consent obtained before any trial related activity and according to local guidelines.

Exclusion Criteria:

1. Postmenopausal women. Postmenopausal status is defined by age>40years with amenorrhea of more than 12 months, associated with serum hormonal levels of the postmenopausal range (either estradiol (E2) < 30 pg/mL and follicle-stimulating hormone (FSH) < 20 mU/mL or E2 ≥ 30 pg/mL and FSH ≥ 20 mU/mL) [30], in the absence of chemotherapy, tamoxifen, or OFS.
2. Patients with primary endocrinal resistance, defined as recurrence within 24 months from the start of adjuvant tamoxifen treatment.
3. Symptomatic and/or life threatening visceral metastases i. Diffuse lymphangitic carcinomatosis. ii. Bulky liver or pulmonary metastases
4. Patients with only non-measurable lesions other than bone metastasis as defined above (e.g., pleural effusion, ascites, etc.).
5. Patients who have received hormonal treatment other than neo/adjuvant tamoxifen

   ± LHRH agonist for their early breast cancer.
6. Patients who received prior chemotherapy for metastatic or recurrent breast cancer.
7. Another malignancy within 5 years prior to enrolment with the exception of adequately treated in-situ carcinoma of the cervix, uterus, basal or squamous cell carcinoma or non-melanomatous skin cancer.
8. Uncontrolled (clinically or radiologically progressive) CNS metastases, carcinomatous meningitis, or leptomeningeal disease.
9. Major surgery within 3 weeks of first study treatment.
10. Chemotherapy, radiotherapy, or other anti-cancer therapy within 2 weeks before randomization. Patients who previously received radiotherapy to 25% of bone marrow are not eligible independent of when it was received.
11. Current treatment with any anti-cancer therapies for advanced disease; any experimental treatment of another clinical trial; therapeutic doses of anticoagulant.

    N.B. Low dose anticoagulants for deep vein thrombosis prophylaxis are allowed. Low molecular weight heparin is allowed. Aspirin is permitted.
12. Active bleeding diathesis.
13. History of non-compliance to medical regimens. Patients unwilling to or unable to comply with the protocol.
14. Pregnant or breast feeding women or those who are not using effective birth control methods. Adequate contraceptives must be used throughout the trial and for 8 weeks after the last study drug administration. Patients must have a negative serum pregnancy test within 7 days prior to first administration of study drug.
15. Prior hematopoietic stem cell or bone marrow transplantation.
16. Current use of food or drugs known to be potent CYP3A4 inhibitors, drugs known to be potent CYP3A4 inducers, and drugs that are known to prolong the QT interval.
17. Known or possible hypersensitivity to goserelin during the adjuvant setting.
18. Any severe and/or uncontrolled medical conditions such as:

    i. Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction < 6months prior to enrollment, serious uncontrolled cardiac arrhythmia ii. Uncontrolled diabetes as defined by fasting serum glucose > 3 x ULN iii. Acute and chronic active infectious disorders (except for Hepatitis B and Hepatitis C positive patients) and non-malignant medical illnesses that are uncontrolled or whose control may be jeopardized by the complications of this study therapy iv. Known human immunodeficiency virus infection v. Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of study drugs (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2019-05-07 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 28 months

SECONDARY OUTCOMES:
Overall response rate | 28 months
Clinical benefit rate | 28 months
Overall survival | 52 months
Incidence of treatment related adverse events | 28 months

CONTACTS AND LOCATIONS:
Locations (1):
- Wits Oncology center, Johannesburg, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Presentation in a conference proceedings in mid 2022 Full publication in January 2023